CLINICAL TRIAL: NCT01891175
Title: Prevention of Maternal Hypotension During Elective Caesarean Section Performed With Spinal Anaesthesia, Through Intermittent Pneumatic Compression System in the Lower Extremities.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Lourdes Trillo, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAESAREANFENI
Record Dates: First submitted 2013-05-24; First posted 2013-07-03 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Hypotension
Keywords: Caesarean; hypotension; Spinal Anaesthesia; intermittent pneumatic compression; lower extremities
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent pneumatic compression (Experimental): With intermittent pneumatic compression of the lower extremities (Covidien / Kendall SCD ™ sequential compression systems) plus phenylephrine perfusion (usual treatment)in elective caesarean section under spinal anaesthesia.
  Interventions: Procedure: Elective caesarean section under spinal anaesthesia.
- Only pheniyephrine perfussion (Active Comparator): No intermittent pneumatic compression of the lower extremities in elective caesarean section under spinal anaesthesia.
  Interventions: Procedure: Elective caesarean section under spinal anaesthesia.

INTERVENTIONS:
Procedure: Elective caesarean section under spinal anaesthesia. — Patients with scheduled caesarean.
  Arms: Intermittent pneumatic compression
Procedure: Elective caesarean section under spinal anaesthesia.
  Arms: Only pheniyephrine perfussion

SUMMARY:
The hypotension defined as 20 % less than the basal SBP (systolic blood pressure)and / or an absolute value <90-100 mmHg, he presents an incident of 80-85% after an anesthesia intradural in the pregnant women, fact that worries for provoking undesirable effects so much in the mother and as in the fetus /newborn baby.

The purpose of this study is to determine the effectiveness of intermittent pneumatic compression system in the lower extremities in order to reduce the vasopressors drugs requirements to maintain hemodynamic stability in pregnant women undergoing elective caesarean sections with an spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years scheduled for elective caesarean section in the third quarter of the pregnancy. Inform Consent signed.

Exclusion Criteria:

* Caesarean section urgent / emergent
* Caesarean section with epidural anaesthesia
* Caesarean section of multiple pregnancies
* Obstetric Pathology: Preeclampsia, Eclampsia, HELLP syndrome (Hemolysis Elevated Liver enzymes Low Platelet count), Small for gestational age (SGA), preterm (<32 weeks)
* Valvular heart disease and / or ischemic
* High blood pressure diagnosed and in treatment.
* Sepsis
* Morbid obesity (BMI> 40)
* Insulin-dependent diabetes
* Block level achieved with spinal anaesthesia> T5
* Patients that can not meet the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The dose of needed vasopressor (phenylephrine). | From the beginning of caesaria section (usually from 32 to 42 weeks of pregnancy) until the end of the surgery.

SECONDARY OUTCOMES:
Effectiveness of Intermittent pneumatic compression system in order to decrease requirements of vasopressors (Phenylephrine). | From the beginning of caesaria section untill discharge of the recovery room ( a maximum of 4 hours).
  Intermittent pneumatic compression system in order to minimise the number of episodes defined as Postoperative nausea and vomiting (POVN) and dizziness associated with hypotension.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Vall d'Hebron Hospital, Barcelona, Barcelona